CLINICAL TRIAL: NCT05550961
Title: APOLLO 11, Consortium of Italian Centers Involved in Treatment of Patients With Lung Cancer Treated With Innovative Therapies: Real World Data and Translational Reaserch
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Politecnico di Milano (Other); Ospedale Policlinico San Martino (Other); Insieme per i Pazienti di Oncologia Polmonare Onlus (IPOP) (Unknown); ASST Grande Ospedale Metropolitano Niguarda (Other); University of Campania Luigi Vanvitelli (Other); Azienda Ospedaliera dei Colli (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); Azienda Ospedaliera "Sant'Andrea" (Other); Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other); IRCCS Sacro Cuore Don Calabria di Negrar (Other); Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other); Istituto Clinico Humanitas (Other); Azienda Unità Sanitaria Locale della Romagna (Other); Istituti Ospitalieri di Cremona (Other)
Responsible Party: Principal Investigator, Arsela Prelaj, Principal Investigator, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT128/22
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: NSCLC; Cancer; Lung Cancer; Adenocarcinoma of Lung; Squamous Cell Lung Cancer
Keywords: #NSCLC; #Immunotherapy; #Targeted Therapy; #Artificial Intelligence
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: About 1000 patients with NSCLC pre-treated with innovative therapy (e.g. immunotherapy, targeted therapy) will be included.
- Prospective Cohort: About 200 patients with NSCLC planned to start an innovative therapy (e.g. immunotherapy, targeted therapy) will be included.

SUMMARY:
APOLLO 11 main aim is to build a strong Italian long-lasting lung cancer network (in around 48 Italian centres) on real world data and translational research by creating a decentralized long-term national database (settle locally in each centre) and a "virtual" multilevel biobank in each centre. Besides, APOLLO 11 will take advantage of the translational research joint effort with the credo "unity is strength".

DETAILED DESCRIPTION:
With the advent of several innovative therapies ("target" therapies, immunotherapy (IO) and/or next generation therapies), the identification of prognostic/predictive and/or resistance biomarkers represents the main goals of translational research in advanced lung cancer (aLC). In particular, with the arrival of IO the treatment landscape of advanced Non-Small Cell Lung Cancer (NSCLC) patients (pts), have radically changed prolonging significantly the overall survival (OS). The role of Programmed Death Ligand 1 (PD-L1) remains undefined and to date no other biomarker are used to select patients for IO. Artificial Intelligence (AI) frameworks, which synthesize and correlate information from different data sources, is a potentially highly efficient instrument to construct algorithms reinforcing the individualized prediction.

APOLLO 11 main aim is to build a strong Italian long-lasting lung cancer network (in around 48 Italian centres) on real world data and translational research by creating a decentralized long-term national database and a "virtual" multilevel biobank. This will allow to avoid worthless dispersion of single institution data, which often remaine unused and inconclusive due to limited number of patients and low statistical power. Besides, APOLLO 11 will take advantage of the translational research joint effort with the credo "unity is strength". The multilevel structure is designed also for smallest centres of give them possibility to contribute to biobank looking at their internal facilities.

APOLLO 11 have the goal to establish the consortium by fully activating at least 20 of the 48 involved centres able to collect data within the database and to guarantee the activation ready for at least 10 biobanks able to collect samples (tumour tissue, blood, stool and urine). Moreover, the key scientific aim of the project is to provide answers about aNSCLC pts treated with IO. In particular, try to find a "software" biomarker able to better predict IO selection compare to standard of care single biomarker (e.g., PD-L1, TMB) using artificial intelligence/machine/deep learning (AI/DL/ML) methodologies. Real world (demographic, histology, PD-L1, molecular, treatment and outcomes information etc), radiomics and where available (from previous researches) multiomic data from all the activated centres will be collected. Furthermore, single-cell RNA sequencing (scRNA seq) analysis will be carry out. Finally, AI/ML/DL will be used to integrate the multisource data, analyse them and develop predictive algorithms of IO efficacy in NSCLC pts. Explainable trustworthy AI (XAI) methodology will be used in order to better understand black box for explaining clinical and biological insight.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent, when applicable, by the patient or legally acceptable representative prior to any mandatory study-specific procedures, sampling, and analyses;
2. Patients must be ≥18 years of age at the time of signing the informed consent;
3. Histologically or cytologically confirmed lung cancer (NSCLC or SCLC) at any stage (I-IV) candidate to receive or already treated with innovative therapies (ICIs, target therapies and next generation therapies).

Exclusion Criteria:

1. Patients who are or will be taking other unapproved antineoplastic therapies concurrently are not eligible.
2. Patients who have not received an oncological systemic innovative therapy at any setting
3. Patients received only local treatments (e.g., only surgery, or only radiotherapy)
4. Patients who received only standard chemotherapy are excluded.
5. Patients who received treatment therapies before 2010 are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC treated with innovative therapies in different Italian Centers will be enrolled in retrospective and prospective cohorts.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Response Rate | About 8 weeks (first radiological evaluation)
  Prediction of response to innovative therapies in NSCLC patients
Progression-Free Survival | From data of enrollment until the date of first documented progression or date of death from any cause, whichever come first, assessed up to 120 months
  Prediction of Progression-Free Survival in NSCLC patients treated with innovative therapies
Overall Survival | From data of enrollment until the date of death from any cause, assessed up to 120 months
  Prediction of Overall Survival in NSCLC patients treated with innovative therapies

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Genova, Principal Investigator — IRCCS Ospedale Policlinico San Martino, Genova; Diego Signorelli, Principal Investigator — ASST Grande Ospedale Metropolitano Niguarda, Milano; Carminia Maria Della Corte, Principal Investigator — Azienda Ospedaliera Universitaria - Università degli Studi della Campania "Luigi Vanvitelli", Napoli; Giuseppe Viscardi, Principal Investigator — Ospedale Monaldi, Azienda Ospedaliera Dei Colli, Monaldi, Napoli; Giulia Galli, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia; Giulio Metro, Principal Investigator — Azienda Ospedaliera Santa Maria della Misercordia, Perugia; Raffaele Giusti, Principal Investigator — Azienda Ospedaliera Univesitaria S. Andrea, Roma; Marianna Macerelli, Principal Investigator — Azienda Ospedaliero-Universitaria Santa Maria Della Misericordia, Udine; Alessandro Inno, Principal Investigator — IRCCS Ospedale sacro Cuore Don Calabria NEGRAR; Rossana Berardi, Principal Investigator — A.O. universitaria Ospedali Riuniti di Ancona; Luca Toschi, Principal Investigator — Fondazione IRCCS Istituto clinico Humanitas; Michela Spreafico, Principal Investigator — Azienda Unità Sanitaria Locale della Romagna, Ravenna; Nicoletta Nanni, Principal Investigator — ASST Ospedale Cremona
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- See also: IPOP website describing APOLLO 11 project — https://www.associazione-ipop.org/progetto-apollo11/

DOCUMENTS (1):
  • Study Protocol (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05550961/Prot_001.pdf